CLINICAL TRIAL: NCT06572891
Title: Compressive Single-piece Implants for Immediate Rehabilitation of Edentulous Maxillectomy Patients with Compromised Ridge: a Study of Patient Satisfaction and Oral Health Related Quality of Life
Brief Title: Compressive Single-piece Implants for Immediate Rehabilitation of Edentulous Maxillectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M0104023RP
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-04

CONDITIONS: Patient Satisfaction
Keywords: VAS; OHIP-EDENT; Obturator Functioning Scale
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional maxillary obturator (Active Comparator): conventional acrylic obturator for each patient
  Interventions: Other: Maxillary obturator
- Implant supported maxillary obturator (Active Comparator): Implant-supported maxillary obturator (compressive implants)
  Interventions: Other: Implant supported obturator

INTERVENTIONS:
Other: Maxillary obturator — conventional acrylic obturator
  Arms: Conventional maxillary obturator
Other: Implant supported obturator — Implants inserted as planned The necks of the implants were bent up to 15 degrees to be parallel.
  * The maxillary obturator was adjusted on the poured mode, modified and access holes will be made above the abutment to be finally relined in the patient mouth at the correct vertical dimension of occlusion to allow for immediate loading protocol.
  * Impressions were made
  Arms: Implant supported maxillary obturator

SUMMARY:
This within-patient study aimed to compare the satisfaction and oral health-related quality of life (OHRQoL) of edentulous maxillectomy patients with and without immediately loaded implant-supported obturator prostheses using single-piece compressive implants.

DETAILED DESCRIPTION:
* Inclusion criteria:

  * Patients with a status eligible for implants after partial or total maxillectomy or partial or total loss of the maxilla.
  * Residual alveolar ridge quantity and quality as verified by cone beam computed tomography (CBCT), especially in the proposed implant sites.
* Exclusion Criteria:

  * Patients with systemic diseases that interfere with surgical implant procedures e.g., uncontrolled diabetes or osteoporosis.
  * Radiation therapy or chemotherapy to the head and neck area (currently or time interval less than 6 months)
  * Patients with local inflammation that may cause interference with implant placement.

All patients were informed about the detailed treatment plan and received a written informed consent to be signed.

II) Preparation of the patient for implant placement:

* Fabrication of maxillary obturator.
* Cone beam computed tomography (CBCT) was performed for all patients to accurately plan implant location, diameter, and angulation.

III) Surgical phase:

* Surgery was performed under local anaesthesia.
* All patients received single-piece compressive implants in the proper positions according to the case demands.
* The patients were prescribed systemic antibiotics for one week, anti-inflammatory, analgesic, and mouthwash.

IV) Prosthetic phase:

* Necks of placed implants bent up to 15 degrees to be parallel placed.
* The maxillary obturator was adjusted on the poured mode, and modified and access holes made above the abutment were finally relined in the patient's mouth at the correct vertical dimension of occlusion to allow for immediate loading protocol.

IV) Evaluation:

* Patient Satisfaction Based on Visual Analog Scale (VAS)
* Oral health impact profile for edentulous patient (OHIP-EDENT)
* Obturator Functioning Scale

ELIGIBILITY:
Inclusion Criteria:

* Patients with a status eligible for implants after partial or total maxillectomy or partial or total loss of the maxilla.
* Residual alveolar ridge quantity and quality will be verified by cone beam computed tomography (CBCT) especially in the proposed implant sites.

Exclusion Criteria:

* Patients with systemic diseases that interfere with surgical implant procedures e.g., uncontrolled diabetes or osteoporosis.
* Radiation therapy or chemotherapy to the head and neck area (currently or time interval less than 6-months)
* Patients with local inflammation that may cause interference with implant placement.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 6 months
  Patient Satisfaction Based on Visual Analog Scale The patients were asked to rate their overall satisfaction with the dentures on a 100-mm visual analogue scale (VAS) for each type of prosthesis. The anchor of the left end of the VAS was defined as 'completely dissatisfied' and that of the opposite side as 'completely satisfied'

SECONDARY OUTCOMES:
Oral health impact profile for edentulous patient (OHIP-EDENT) | 6 months
  Oral health impact profile for edentulous patients (OHIP-EDENT). The total 19 items are defined to measure seven domains: (1) functional limitation (3 items), (2) pain (4 items), (3) psychological discomfort (2 items), (4) physical disability (3 items), (5) psychological disability (2 items), (6) social disability (3 items), and (7) handicap(2 items). Each item is scored on a Likert scale from 1 ('Never') to 5 ('Very often'). The outcomes of the OHIP-EDENT can have ranged from 19 to 95. A score of 19 means that dental problems do not affect daily life at all, whereas a score of 95 means that dental problems affect daily life very often.
- Obturator Functioning Scale | 6 months
  Obturator functioning scale was assessed in 1-15 questions in terms of no difficulty on a 5-point Likert Scale. Points 1 represent "not at all difficult" and point 2 stood for "a little difficult". Point 1 and 2 were considered as "No Difficulty" on the scale. Points 3, stood for 'somewhat difficult', point 4 for 'very much difficult' and point 5 for 'extremely difficult' and point 3, 4, and 5 were considered as 'Difficulty'.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No